CLINICAL TRIAL: NCT00970307
Title: Immunogenicity and Safety Study of GlaxoSmithKline Biologicals' GSK2202083A Vaccine in Healthy Infants at 2, 3 and 4 Months of Age
Brief Title: Immunogenicity and Safety Study of GSK Biologicals' GSK2202083A Vaccine in Healthy Infants at 2, 3 and 4 Months of Age
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 112157; 2009-010431-41 (EudraCT Number)
Record Dates: First submitted 2009-08-27; First posted 2009-09-02 (Estimated); Results first posted 2017-04-14 (Actual); Last update posted 2020-01-03 (Actual); Status verified 2019-12

CONDITIONS: Tetanus; Diphtheria; Haemophilus Influenzae Type b; Poliomyelitis; Acellular Pertussis; Hepatitis B; Diphtheria-Tetanus-aPertussis-Hepatitis B-Poliomyelitis-Haemophilus Influenzae Type b-Neisseria Meni
MeSH Terms: conditions — Tetanus; Diphtheria; Haemophilus Infections; Poliomyelitis; Hepatitis B | interventions — 10-valent pneumococcal vaccine; diphtheria-tetanus-acellular pertussis-inactivated poliovirus-Haemophilus influenzae b conjugate-hepatitis B vaccine

ARMS (3):
- GSK2202083A + SYNFLORIX GROUP (Experimental): Healthy male and female infants between and including 8 to 12 weeks at the time of the first vaccination, who received 3 doses of GSK2202083A vaccine and Synflorix™ vaccine at 2, 3 and 4 months of age and 2 doses of Rotarix™ vaccine at 2 and 3 months of age. GSK2202083A and Synflorix™ vaccines were administered intramuscularly into the right and left thigh, while Rotarix™ vaccine was administered orally.
  Interventions: Biological: GSK2202083A vaccine; Biological: 10-valent pneumococcal vaccine (GSK 1024850A)
- INFANRIX HEXA + MENJUGATE GROUP (Active Comparator): Healthy male and female infants between and including 8 to 12 weeks at the time of the first vaccination, who received 3 doses of Infanrix hexa™ vaccine at 2, 3 and 4 months of age, 2 doses of Menjugate® vaccine at 3 and 4 months of age and 2 doses of Rotarix™ vaccine at 2 and 3 months of age. Infanrix hexa™ and Menjugate® vaccines were administered intramuscularly into the right and left thigh, while Rotarix™ vaccine was administered orally.
  Interventions: Biological: Infanrix hexa™; Biological: Menjugate®
- INFANRIX HEXA + SYNFLORIX GROUP (Active Comparator): Healthy male and female infants between and including 8 to 12 weeks at the time of the first vaccination, who received 3 doses of Infanrix hexa™ vaccine and Synflorix™ vaccine at 2, 3 and 4 months of age and 2 doses of Rotarix™ vaccine at 2 and 3 months of age. Infanrix hexa™ and Synflorix™ vaccines were administered intramuscularly into the right and left thigh, while Rotarix™ vaccine was administered orally.
  Interventions: Biological: 10-valent pneumococcal vaccine (GSK 1024850A); Biological: Infanrix hexa™

INTERVENTIONS:
Biological: GSK2202083A vaccine — Intramuscular, three doses
  Arms: GSK2202083A + SYNFLORIX GROUP
Biological: 10-valent pneumococcal vaccine (GSK 1024850A) — Intramuscular, three doses
  Arms: GSK2202083A + SYNFLORIX GROUP; INFANRIX HEXA + SYNFLORIX GROUP
Biological: Infanrix hexa™ — Intramuscular, three doses
  Arms: INFANRIX HEXA + MENJUGATE GROUP; INFANRIX HEXA + SYNFLORIX GROUP
Biological: Menjugate® — Intramuscular, two doses
  Arms: INFANRIX HEXA + MENJUGATE GROUP

SUMMARY:
This study will evaluate the safety and immunogenicity of GSK Biologicals' GSK2202083A vaccine co-administered with GSK Biologicals' 10-valent pneumococcal conjugate (GSK1024850A) vaccine given as a three-dose primary vaccination course at 2, 3 and 4 months of age.

DETAILED DESCRIPTION:
In accordance with the local recommended immunisation schedule, all subjects will receive 2 doses of GSK Biologicals' Human Rotavirus Vaccine (Rotarix) at 2 and 3 months of age.

ELIGIBILITY:
Inclusion Criteria:

* A male or female infant between, and including, 8 and 12 weeks of age at the time of the first vaccination.
* Born after a gestation period of 36 to 42 weeks inclusive.
* Subjects should have received one dose of hepatitis B vaccination at birth as per local recommendations.
* Subjects who the investigator believes that their parent(s)/LAR can and will comply with the requirements of the protocol.
* Written informed consent obtained from the parent/LAR of the subject.
* Healthy subjects as established by medical history and clinical examination before entering into the study.

Exclusion Criteria:

* Use of any investigational or non-registered product other than the study vaccines within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Chronic administration of immunosuppressants or other immune-modifying drugs since birth.
* Administration of immunoglobulins and/or any blood products since birth or planned administration during the study period.
* Administration of any vaccine since birth, with exception of HBV and Bacillus Calmette-Guérin, or planned administration during the study period.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product.
* Evidence of previous or intercurrent diphtheria, tetanus, pertussis, hepatitis B, polio, Hib, pneumococcal and/or MenC disease.
* History of seizures or progressive neurological disease.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccines.
* Major congenital defects or serious chronic illness.

The following condition is temporary or self-limiting, and a subject may be vaccinated once the condition has resolved if no other exclusion criteria is met:

• Current febrile illness or axillary temperature >= 38.5 ºC or other moderate to severe illness within 24 hours of study vaccine administration.

Ages: 8 Weeks to 12 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 421 (Actual)
Dates: Start 2009-08-13 (Actual); Primary Completion 2010-01-27 (Actual); Study Completion 2010-01-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (8):
- Poland (8):
  - GSK Investigational Site, Bydgoszcz
  - GSK Investigational Site, Dębica
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Siemianowice Śląskie
  - GSK Investigational Site, Tarnów
  - GSK Investigational Site, Torun
  - GSK Investigational Site, Trzebnica
  - GSK Investigational Site, Wroclaw

IPD SHARING:
Plan to Share IPD: Yes
IPD is available via the Clinical Study Data Request site (click on the link provided below)
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=136

REFERENCES:
- [Background] Szenborn L, Czajka H, Brzostek J, Konior R, Caubet M, Ulianov L, Leyssen M. A randomized, controlled trial to assess the immunogenicity and safety of a heptavalent diphtheria, tetanus, pertussis, hepatitis B, poliomyelitis, hib and meningococcal serogroup C combination vaccine administered at 2, 3, 4 and 12-18 months of age. Pediatr Infect Dis J. 2013 Jul;32(7):777-85. doi: 10.1097/INF.0b013e31828d6b20. PMID 23838777
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 112157 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 112157 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 112157 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 112157 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 112157 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 112157 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 112157 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: During the screening the following steps occurred: check for inclusion/exclusion criteria, contraindications/precautions, medical history of the subjects and signing informed consent forms.
Period: Overall Study
Arm/Group | GSK2202083A + Synflorix Group | Infanrix Hexa + Menjugate Group | Infanrix Hexa + Synflorix Group
Started | 141 | 139 | 141
Completed | 138 | 136 | 139
Not Completed | 3 | 3 | 2
Not completed — Serious Adverse Event | 1 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK2202083A + Synflorix Group | Infanrix Hexa + Menjugate Group | Infanrix Hexa + Synflorix Group | Total
Number analyzed (Participants) | 141 | 139 | 141 | 421
Age, Continuous [Mean (Standard Deviation); unit: Weeks] | 8.5 (0.98) | 8.7 (1.02) | 8.7 (1.13) | 8.63 (1.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74 | 86 | 68 | 228
  Male | 67 | 53 | 73 | 193
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White-Caucasian/European heritage | 141 | 139 | 141 | 421

OUTCOME MEASURES:

1. Primary Outcome: Number of Seroprotected Subjects Against Polyribosyl-Ribitol-Phosphate (PRP)
Description: A seroprotected subject was defined as a subject with anti-PRP antibody concentrations greater than or equal to (≥) 0.15 micrograms per milliliter (µg/mL).
Time Frame: At Month 3
Population: The analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity, which included all evaluable subjects for whom immunogenicity data and assay results were available for antibodies against at least one study vaccine antigen component at the post-primary vaccination blood-sampling time point.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2202083A + Synflorix Group | Infanrix Hexa + Menjugate Group | Infanrix Hexa + Synflorix Group
Number analyzed (Participants) | 126 | 132 | 131
Participants | 126 | 123 | 130
Statistical Analysis 1: Comparison: GSK2202083A + Synflorix Group vs Infanrix Hexa + Synflorix Group; Test type: Non-Inferiority — Criterion for evaluation of Non-inferiority: the upper limit of Standardised asymptotic 95% confidence interval lower or equal to 10%; Difference in percentage = -0.76, 95% CI 2-sided [-4.21 to 2.22]

2. Primary Outcome: Number of Seroprotected Subjects Against Neisseria Meningitidis Serogroup C Using Baby Rabbit Complement (rSBA-MenC)
Description: A seroprotected subject was defined as a subject with rSBA-MenC titers greater than or equal to (≥) 1:8.
Time Frame: At Month 3
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2202083A + Synflorix Group | Infanrix Hexa + Menjugate Group | Infanrix Hexa + Synflorix Group
Number analyzed (Participants) | 126 | 130 | 128
Participants | 124 | 127 | 10
Statistical Analysis 1: Comparison: GSK2202083A + Synflorix Group vs Infanrix Hexa + Menjugate Group; Test type: Non-Inferiority — Criterion for evaluation of Non-inferiority: the upper limit of Standardized asymptotic 95% confidence interval lower or equal to 10%; Difference in percentage = -0.72, 95% CI 2-sided [-5.19 to 3.57]

3. Secondary Outcome: Anti-PRP Antibody Concentrations
Description: Concentrations were expressed as geometric mean concentrations (GMCs) for the seroprotection cut-off value of ≥ 0.15 µg/mL.
Time Frame: At Months 0 and 3
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | GSK2202083A + Synflorix Group | Infanrix Hexa + Menjugate Group | Infanrix Hexa + Synflorix Group
Number analyzed (Participants) | 126 | 132 | 131
µg/mL
  Anti-PRP, Month 0: number analyzed (Participants) | 124 | 127 | 127
  Anti-PRP, Month 0 | 0.197 [0.162 to 0.24] | 0.152 [0.125 to 0.184] | 0.176 [0.143 to 0.217]
  Anti-PRP, Month 3 | 4.255 [3.591 to 5.043] | 1.123 [0.89 to 1.416] | 1.721 [1.383 to 2.143]

4. Secondary Outcome: Antibody Titers Against rSBA-MenC
Description: The seroprotection cut-off value of the assay was an antibody titer ≥ 1:8.
Time Frame: At Months 0 and 3
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | GSK2202083A + Synflorix Group | Infanrix Hexa + Menjugate Group | Infanrix Hexa + Synflorix Group
Number analyzed (Participants) | 126 | 130 | 128
Titers
  rSBA-MenC, Month 0: number analyzed (Participants) | 118 | 119 | 120
  rSBA-MenC, Month 0 | 4.3 [4 to 4.7] | 4.8 [4.2 to 5.5] | 4.2 [4 to 4.5]
  rSBA-MenC, Month 3 | 786.9 [637.2 to 971.9] | 2674 [2125.1 to 3364.7] | 6.1 [4.7 to 8]

5. Secondary Outcome: Number of Seropositive Subjects for Anti-polysaccharide Neisseria Meningitidis Serogroup C (Anti-PSC)
Description: A seropositive subject was defined as a subject with anti-PSC antibody concentration ≥ 0.3 µg/mL.
Time Frame: At Month 3
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2202083A + Synflorix Group | Infanrix Hexa + Menjugate Group | Infanrix Hexa + Synflorix Group
Number analyzed (Participants) | 125 | 126 | 132
Participants | 124 | 125 | 8

6. Secondary Outcome: Anti-PSC Antibody Concentrations
Description: Concentrations were expressed as geometric mean concentrations (GMCs) for the seropositivity cut-off value of ≥ 0.3 µg/mL.
Time Frame: At Months 0 and 3
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | GSK2202083A + Synflorix Group | Infanrix Hexa + Menjugate Group | Infanrix Hexa + Synflorix Group
Number analyzed (Participants) | 125 | 126 | 132
µg/mL
  Anti-PSC, Month 0: number analyzed (Participants) | 122 | 121 | 126
  Anti-PSC, Month 0 | 0.17 [0.16 to 0.19] | 0.17 [0.16 to 0.19] | 0.18 [0.16 to 0.2]
  Anti-PSC, Month 3 | 19.15 [16.88 to 21.74] | 18.1 [15.91 to 20.59] | 0.19 [0.16 to 0.22]

7. Secondary Outcome: Number of Seroprotected Subjects Against Diphtheria (D) and Tetanus (T)
Description: A seroprotected subject was defined as a subject with anti-D or anti-T antibody concentrations ≥ 0.1 international units per milliliter (IU/mL).
Time Frame: At Month 3
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2202083A + Synflorix Group | Infanrix Hexa + Menjugate Group | Infanrix Hexa + Synflorix Group
Number analyzed (Participants) | 126 | 132 | 132
Participants
  Anti-D | 126 | 132 | 132
  Anti-T | 126 | 132 | 132

8. Secondary Outcome: Anti-D and Anti-T Antibody Concentrations
Description: Concentrations were expressed as geometric mean concentrations (GMCs) for the seroprotection cut-off value of ≥ 0.1 IU/mL.
Time Frame: At Month 3
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | GSK2202083A + Synflorix Group | Infanrix Hexa + Menjugate Group | Infanrix Hexa + Synflorix Group
Number analyzed (Participants) | 126 | 132 | 132
IU/mL
  Anti-D | 1.671 [1.471 to 1.899] | 1.437 [1.286 to 1.606] | 1.421 [1.270 to 1.591]
  Anti-T | 3.966 [3.65 to 4.309] | 1.595 [1.422 to 1.79] | 2.458 [2.198 to 2.75]

9. Secondary Outcome: Number of Seropositive Subjects for Anti-pertussis Toxoid (Anti-PT), Anti-filamentous Haemagglutinin (Anti-FHA) and Anti-pertactin (Anti-PRN)
Description: A seropositive subject was defined as a subject with anti-PT, anti-FHA or anti-PRN concentrations ≥ 5 enzyme-linked immunosorbent assay (ELISA) units per milliliter (EL.U/mL).
Time Frame: At Month 3
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2202083A + Synflorix Group | Infanrix Hexa + Menjugate Group | Infanrix Hexa + Synflorix Group
Number analyzed (Participants) | 127 | 132 | 132
Participants
  Anti-PT | 127 | 132 | 132
  Anti-FHA: number analyzed (Participants) | 127 | 131 | 132
  Anti-FHA | 127 | 131 | 132
  Anti-PRN: number analyzed (Participants) | 126 | 132 | 131
  Anti-PRN | 126 | 132 | 131

10. Secondary Outcome: Anti-PT, Anti-FHA and Anti-PRN Antibody Concentrations
Description: Concentrations were expressed as geometric mean concentrations (GMCs) for the seropositivity cut-off value of ≥ 5 EL.U/mL.
Time Frame: At Months 0 and 3
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | GSK2202083A + Synflorix Group | Infanrix Hexa + Menjugate Group | Infanrix Hexa + Synflorix Group
Number analyzed (Participants) | 127 | 132 | 132
EL.U/mL
  Anti-PT, Month 0: number analyzed (Participants) | 123 | 129 | 129
  Anti-PT, Month 0 | 3.5 [3.1 to 4] | 3.6 [3.1 to 4] | 3.8 [3.3 to 4.4]
  Anti-PT, Month 3 | 36.1 [32.8 to 39.8] | 41.7 [37.4 to 46.4] | 37.6 [34.2 to 41.4]
  Anti-FHA, Month 0: number analyzed (Participants) | 125 | 130 | 127
  Anti-FHA, Month 0 | 12.9 [10.7 to 15.6] | 11.9 [9.5 to 14.9] | 13.2 [10.6 to 16.5]
  Anti-FHA, Month 3: number analyzed (Participants) | 127 | 131 | 132
  Anti-FHA, Month 3 | 110.9 [98.1 to 125.4] | 136.4 [121.3 to 153.5] | 112.7 [100.9 to 126]
  Anti-PRN, Month 0: number analyzed (Participants) | 127 | 131 | 132
  Anti-PRN, Month 0 | 5.3 [4.4 to 6.4] | 4.3 [3.7 to 5.1] | 5.4 [4.5 to 6.5]
  Anti-PRN, Month 3: number analyzed (Participants) | 126 | 132 | 131
  Anti-PRN, Month 3 | 70.3 [59.6 to 82.8] | 107.4 [93 to 124.2] | 90.4 [78.1 to 104.6]

11. Secondary Outcome: Number of Subjects With a Vaccine Response to Anti-PT, Anti-FHA and Anti-PRN
Description: A subject with a vaccine response was defined as either an initially seronegative subject with anti-PT, anti-FHA or anti-PRN concentrations ≥ 5 EL.U/mL or an initially seropositive subjects with antibody concentrations one month after the primary vaccination ≥ 1 fold the-pre vaccination antibody concentration.
Time Frame: At Month 3
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2202083A + Synflorix Group | Infanrix Hexa + Menjugate Group | Infanrix Hexa + Synflorix Group
Number analyzed (Participants) | 126 | 131 | 131
Participants
  Anti-PT: number analyzed (Participants) | 123 | 129 | 129
  Anti-PT | 121 | 124 | 122
  Anti-FHA: number analyzed (Participants) | 125 | 129 | 127
  Anti-FHA | 116 | 123 | 120
  Anti-PRN | 112 | 123 | 123

12. Secondary Outcome: Number of Seroprotected and Seropositive Subjects for Anti-hepatitis B Surface Antigen (Anti-HBs)
Description: A seroprotected subject was defined as a subject with anti-HBs antibody concentrations ≥ 10 mIU/mL. A seropositive subject was defined as a subjects with anti-HBs antibody concentrations ≥ 3.3 mIU/mL. A decrease in the specificity of the anti-HB ELISA had been observed in some studies for low levels of antibody (10-100 mIU/mL). All the available blood samples initially tested with ELISA were re-tested using the Chemi Luminescence Immuno Assay (CLIA) approved by the US Food and Drug Administration (FDA). The table shows updated results following partial or complete retesting/reanalysis.
Time Frame: At Month 3
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2202083A + Synflorix Group | Infanrix Hexa + Menjugate Group | Infanrix Hexa + Synflorix Group
Number analyzed (Participants) | 116 | 124 | 122
Participants
  Anti-HBs ≥ 10 mIU/mL | 116 | 124 | 122
  Anti-HBs ≥ 3.3 mIU/mL | 116 | 124 | 122

13. Secondary Outcome: Anti-HBs Antibody Concentrations
Description: Antibody concentrations were expressed as GMCs. The seroprotection cut-off used was of ≥ 10 mIU/mL. A decrease in the specificity of the anti-HB ELISA had been observed in some studies for low levels of antibody (10-100 mIU/mL). All the available blood samples initially tested with ELISA were re-tested using the CLIA approved by the FDA. The table shows updated results following partial or complete retesting/reanalysis.
Time Frame: At Month 3
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | GSK2202083A + Synflorix Group | Infanrix Hexa + Menjugate Group | Infanrix Hexa + Synflorix Group
Number analyzed (Participants) | 116 | 124 | 122
mIU/mL | 1001.4 [826.1 to 1213.9] | 1187.7 [997.8 to 1413.7] | 1073.2 [886.3 to 1299.5]

14. Secondary Outcome: Number of Seroprotected Subjects for Anti-poliovirus (Anti-polio) Types 1, 2 and 3
Description: A seroprotected subject was defined as a subject with anti-polio type 1, 2 or 3 antibody titers ≥ 1:8.
Time Frame: At Month 3
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2202083A + Synflorix Group | Infanrix Hexa + Menjugate Group | Infanrix Hexa + Synflorix Group
Number analyzed (Participants) | 91 | 103 | 92
Participants
  Anti-polio type 1 | 91 | 103 | 92
  Anti-polio type 2 | 90 | 101 | 91
  Anti-polio type 3: number analyzed (Participants) | 90 | 102 | 91
  Anti-polio type 3 | 90 | 102 | 91

15. Secondary Outcome: Anti-polio Types 1, 2 and 3 Antibody Titers
Description: Titers were expressed as geometric mean titers (GMTs) for the seroprotection cut-off value of ≥ 1:8.
Time Frame: At Month 3
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | GSK2202083A + Synflorix Group | Infanrix Hexa + Menjugate Group | Infanrix Hexa + Synflorix Group
Number analyzed (Participants) | 91 | 103 | 92
Titers
  Anti-polio type 1 | 132.3 [104.7 to 167.3] | 156.7 [127.2 to 193] | 126.2 [98.9 to 161]
  Anti-polio type 2 | 97.4 [74 to 128.1] | 104.3 [80.8 to 134.7] | 95.8 [74.4 to 123.3]
  Anti-polio type 3: number analyzed (Participants) | 90 | 102 | 91
  Anti-polio type 3 | 275.6 [218.2 to 348.1] | 313.1 [250.7 to 391] | 257.1 [203.8 to 324.3]

16. Secondary Outcome: Number of Seropositive Subjects for Anti-pneumococcal (Anti-pneumo) Serotypes
Description: A seropositive subject was defined as a subject with anti-pneumo concentrations ≥ 0.05 µg/mL. The anti-pneumo serotypes assessed were: 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F.
Time Frame: At Month 3
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2202083A + Synflorix Group | Infanrix Hexa + Menjugate Group | Infanrix Hexa + Synflorix Group
Number analyzed (Participants) | 127 | 127 | 129
Participants
  Anti-pneumo 1: number analyzed (Participants) | 125 | 123 | 125
  Anti-pneumo 1 | 125 | 37 | 124
  Anti-pneumo 4: number analyzed (Participants) | 122 | 119 | 128
  Anti-pneumo 4 | 122 | 21 | 127
  Anti-pneumo 5: number analyzed (Participants) | 126 | 111 | 127
  Anti-pneumo 5 | 126 | 44 | 126
  Anti-pneumo 6B: number analyzed (Participants) | 119 | 120 | 126
  Anti-pneumo 6B | 114 | 28 | 117
  Anti-pneumo 7F: number analyzed (Participants) | 125 | 123 | 129
  Anti-pneumo 7F | 125 | 56 | 128
  Anti-pneumo 9V: number analyzed (Participants) | 126 | 121 | 127
  Anti-pneumo 9V | 126 | 37 | 126
  Anti-pneumo 14: number analyzed (Participants) | 126 | 119 | 128
  Anti-pneumo 14 | 126 | 106 | 128
  Anti-pneumo 18C: number analyzed (Participants) | 122 | 111 | 126
  Anti-pneumo 18C | 122 | 52 | 126
  Anti-pneumo 19F: number analyzed (Participants) | 127 | 121 | 128
  Anti-pneumo 19F | 127 | 88 | 127
  Anti-pneumo 23F: number analyzed (Participants) | 126 | 127 | 129
  Anti-pneumo 23F | 123 | 34 | 124

17. Secondary Outcome: Anti-pneumo Antibody Concentrations
Description: Concentrations were expressed as geometric mean concentrations (GMCs) for the seropositivity cut-off value of ≥ 0.05 µg/mL.
Time Frame: At Month 3
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | GSK2202083A + Synflorix Group | Infanrix Hexa + Menjugate Group | Infanrix Hexa + Synflorix Group
Number analyzed (Participants) | 127 | 127 | 129
µg/mL
  Anti-pneumo 1: number analyzed (Participants) | 125 | 123 | 125
  Anti-pneumo 1 | 1.53 [1.36 to 1.72] | 0.04 [0.04 to 0.05] | 1.41 [1.2 to 1.65]
  Anti-pneumo 4: number analyzed (Participants) | 122 | 119 | 128
  Anti-pneumo 4 | 1.92 [1.66 to 2.22] | 0.04 [0.03 to 0.04] | 1.99 [1.69 to 2.33]
  Anti-pneumo 5: number analyzed (Participants) | 126 | 111 | 127
  Anti-pneumo 5 | 2.23 [1.99 to 2.5] | 0.05 [0.04 to 0.06] | 2.23 [1.9 to 2.61]
  Anti-pneumo 6B: number analyzed (Participants) | 119 | 120 | 126
  Anti-pneumo 6B | 0.4 [0.32 to 0.49] | 0.04 [0.03 to 0.04] | 0.44 [0.35 to 0.55]
  Anti-pneumo 7F: number analyzed (Participants) | 125 | 123 | 129
  Anti-pneumo 7F | 2.26 [2.02 to 2.53] | 0.06 [0.05 to 0.07] | 2.24 [1.95 to 2.56]
  Anti-pneumo 9V: number analyzed (Participants) | 126 | 121 | 127
  Anti-pneumo 9V | 2.16 [1.9 to 2.46] | 0.05 [0.04 to 0.06] | 1.99 [1.72 to 2.3]
  Anti-pneumo 14: number analyzed (Participants) | 126 | 119 | 128
  Anti-pneumo 14 | 3.75 [3.23 to 4.36] | 0.22 [0.17 to 0.28] | 3.75 [3.26 to 4.32]
  Anti-pneumo 18C: number analyzed (Participants) | 122 | 111 | 126
  Anti-pneumo 18C | 3.83 [3.22 to 4.56] | 0.05 [0.04 to 0.07] | 2.51 [2.11 to 2.99]
  Anti-pneumo 19F: number analyzed (Participants) | 127 | 121 | 128
  Anti-pneumo 19F | 3.99 [3.37 to 4.72] | 0.1 [0.08 to 0.13] | 3.86 [3.19 to 4.66]
  Anti-pneumo 23F: number analyzed (Participants) | 126 | 127 | 129
  Anti-pneumo 23F | 0.68 [0.55 to 0.84] | 0.04 [0.03 to 0.05] | 0.63 [0.5 to 0.79]

18. Secondary Outcome: Number of Seropositive Subjects for Anti-protein D (Anti-PD)
Description: A seropositive subject was defined as a subject with anti-PD concentrations ≥ 100 EL.U/mL.
Time Frame: At Month 3
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2202083A + Synflorix Group | Infanrix Hexa + Menjugate Group | Infanrix Hexa + Synflorix Group
Number analyzed (Participants) | 126 | 129 | 131
Participants | 126 | 18 | 130

19. Secondary Outcome: Anti-PD Antibody Concentrations
Description: Concentrations were expressed as geometric mean concentrations (GMCs) for the seropositivity cut-off value of ≥ 100 EL.U/mL.
Time Frame: At Month 3
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | GSK2202083A + Synflorix Group | Infanrix Hexa + Menjugate Group | Infanrix Hexa + Synflorix Group
Number analyzed (Participants) | 126 | 129 | 131
EL.U/mL | 1622.8 [1433.4 to 1837.1] | 63.3 [56.3 to 71.2] | 1561.6 [1359.2 to 1794]

20. Secondary Outcome: Number of Subjects With Any Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = incidence of a local symptom irrespective of intensity grade.
Time Frame: During the 8-day (Days 0-7) post-vaccination period after any vaccination
Population: The analysis was performed on the Total Vaccinated Cohort, which included all vaccinated subjects for whom data were available and had the symptom sheets filled in.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2202083A + Synflorix Group | Infanrix Hexa + Menjugate Group | Infanrix Hexa + Synflorix Group
Number analyzed (Participants) | 140 | 138 | 141
Participants
  Any pain | 66 | 70 | 85
  Any redness | 83 | 81 | 83
  Any swelling | 64 | 50 | 71

21. Secondary Outcome: Number of Subjects With Any Solicited General Symptoms
Description: Assessed solicited general symptoms were drowsiness, irritability, loss of appetite and fever (defined as axillary temperature ≥ 37.5°C). Any= incidence of a general symptom irrespective of intensity grade and relationship to vaccination.
Time Frame: During the 8-day (Days 0-7) post-vaccination period after any vaccination
Population: as for outcome 20
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2202083A + Synflorix Group | Infanrix Hexa + Menjugate Group | Infanrix Hexa + Synflorix Group
Number analyzed (Participants) | 140 | 138 | 141
Participants
  Any drowsiness | 105 | 91 | 107
  Any irritability | 108 | 101 | 113
  Any loss of appetite | 72 | 62 | 72
  Any fever | 53 | 38 | 61

22. Secondary Outcome: Number of Subjects With Unsolicited Adverse Events (AEs)
Description: An unsolicited AE was any AE (i.e. any untoward medical occurrence in a patient or clinical investigation subject, temporally associated with use of a medicinal product, whether or not considered related to the medicinal product) reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms.
Time Frame: During the 31-day (Days 0-30) post-vaccination period after any vaccination
Population: The analysis was performed on the Total Vaccinated Cohort, which included all vaccinated subjects for whom data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2202083A + Synflorix Group | Infanrix Hexa + Menjugate Group | Infanrix Hexa + Synflorix Group
Number analyzed (Participants) | 141 | 139 | 141
Participants | 61 | 52 | 61

23. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: SAEs were defined as medical occurrences that resulted in death, were life threatening, required hospitalization or prolongation of hospitalization or resulted in disability/incapacity.
Time Frame: During the entire study period (from Month 0 to Month 3)
Population: as for outcome 22
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2202083A + Synflorix Group | Infanrix Hexa + Menjugate Group | Infanrix Hexa + Synflorix Group
Number analyzed (Participants) | 141 | 139 | 141
Participants | 5 | 6 | 3

ADVERSE EVENTS:
Time Frame: Solicited local and general symptoms: during the 8-day (Days 0-7) post-vaccination period. Unsolicited adverse events: during the 31-day (Days 0-30) post-vaccination. Serious adverse events: during the entire study period (from Month 0 up to Month 3).
Arm/Group | GSK2202083A + Synflorix Group | Infanrix Hexa + Menjugate Group | Infanrix Hexa + Synflorix Group
All-Cause Mortality (participants affected / at risk) | 0/141 | 0/139 | 0/141
Serious Adverse Events (participants affected / at risk) | 5/141 | 6/139 | 3/141
Other Adverse Events (participants affected / at risk) | 130/141 | 129/139 | 137/141
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GSK2202083A + Synflorix Group (N=141) | Infanrix Hexa + Menjugate Group (N=139) | Infanrix Hexa + Synflorix Group (N=141)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1
Bronchopneumonia (Infections and infestations) | 2 | 1 | 0
Bronchitis (Infections and infestations) | 1 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 1 | 0
Bronchiolitis (Infections and infestations) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1
Otitis media (Infections and infestations) | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GSK2202083A + Synflorix Group (N=141) | Infanrix Hexa + Menjugate Group (N=139) | Infanrix Hexa + Synflorix Group (N=141)
Pain (General disorders) | 66 | 70 | 85
Redness (General disorders) | 83 | 81 | 83
Swelling (General disorders) | 64 | 50 | 71
Drowsiness (General disorders) | 105 | 91 | 107
Irritability (General disorders) | 108 | 101 | 113
Loss of appetite (General disorders) | 72 | 62 | 72
Temperature (Axillary) (General disorders) | 53 | 38 | 61
Rhinitis (Infections and infestations) | 11 | 18 | 17
Upper respiratory tract infection (Infections and infestations) | 10 | 7 | 10
Nasopharyngitis (Infections and infestations) | 9 | 4 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.